CLINICAL TRIAL: NCT01485874
Title: A Phase I-II Clinical Trial of Pegylated Liposomal Doxorubicin (Doxil®) in Combination With BIBF 1120 in Patients With Ovarian Cancer: Hoosier Oncology Group GYN10-149
Brief Title: Doxorubicin + BIBF 1120 in Patients for Ovarian Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding withdrawn due to drug unavailability
Sponsor: Hoosier Cancer Research Network (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GYN10-149
Record Dates: First submitted 2011-12-02; First posted 2011-12-06 (Estimated); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Ovarian Cancer
Keywords: BIBF 1120
MeSH Terms: conditions — Ovarian Neoplasms | interventions — liposomal doxorubicin; nintedanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Doxil + BIBF 1120 (Experimental)
  Interventions: Drug: Doxil (Pegylated Liposomal Doxorubicin); Drug: BIBF 1120

INTERVENTIONS:
Drug: Doxil (Pegylated Liposomal Doxorubicin) — Phases I and II: 40 mg/m2 IV over 60 min (+/- 15 min) on day 1 of 28-day cycle
Drug: BIBF 1120 — Phase I: Escalating cohorts days -2 through +2, orally 100mg bid, 150mg bid, 200mg bid
  Phase II: MTD orally, bid, day 2 of 28-day cycle

SUMMARY:
The purpose of this trial is to determine whether BIBF 1120 can be safely combined with pegylated liposomal doxorubicin (phase I), and to determine the clinical activity of the combination in patients with platinum-resistant ovarian cancer (phase II).

DETAILED DESCRIPTION:
OUTLINE: This is a phase I/II multi-center study.

Phase I:

All patients will receive a fixed dose of pegylated liposomal doxorubicin (Doxil) of 40 mg/m2 administered IV every 28 days. The dose of BIBF 1120 will be escalated in successive cohorts of patients. A maximum of 12 cycles of combined therapy will be administered corresponding to maximum cumulative dose of PLD of 480 mg/m2. Continuation therapy with single agent BIBF 1120 may continue for selected patients.

The escalation phase will follow the standard 3+3 design. Patients will be accrued to each dose level in cohorts of up to 3-6 evaluable patients. Escalation will continue until a DLT is observed, the highest dose level is reached, or medical judgment indicates. An expansion cohort of 3 to 6 patients will be treated at the MTD (or highest dose level if the MTD is not reached), in order to ensure tolerability of the regimen prior to initiating the Phase II component of the study.

Phase II:

Patients will receive a fixed dose of pegylated liposomal doxorubicin (Doxil) of 40 mg/m2 administered IV every 28 days. Patients will be treated at either dose Level +2 or the MTD dose level of BIBF 1120 as defined by the Phase I cohort. Each cycle will be 28 days. Patients will continue treatment with the combination therapy for a total of up to 12 cycles.

ECOG Performance Status 0-1

Life Expectancy: Not specified

Hematopoietic:

* Absolute neutrophil count ≥ 1500 cells/mm3
* White cell blood count ≥ 3000 cells/mm3
* Hemoglobin ≥ 9.0 g/dL (can be post-transfusion)
* Platelets ≥ 100,000/mm3 (can not be post-transfusion)

Hepatic:

* Aspartate aminotransferase and alanine aminotransferase less than or equal to 2.5 times upper limit of normal (ULN)
* Total serum bilirubin ≤ 1.5 times ULN
* Alkaline phosphatase ≤ 2.5 times ULN

Renal:

* Creatinine levels ≤ 1.5 times ULN

Cardiovascular:

* Baseline left ventricular ejection fraction greater than 50%
* International Normalized ratio(INR) ≤ 1.5 times ULN, except patients on stable doses of coumadin or low molecular weight heparin NOTE: Patients on stable doses of coumadin or low molecular weight heparin are eligible if anticoagulant doses have been stable and no bleeding complications were recorded.
* Partial thromboplastin time (PTT) ≤1.5 times ULN

This study was terminated due to drug availability and Phase II never opened.

ELIGIBILITY:
Inclusion Criteria:

* Platinum-resistant (recurrence within 6 months of a platinum-containing regimen) or platinum refractory (progression while on platinum) disease.
* Measurable disease as defined by RECIST v1.1 criteria on screening testing
* Be ≥18 years of age at the time of providing written informed consent for participation.
* Give written, informed consent for participation in the protocol.
* Must consent to correlative blood sample collections.
* Be at least 4 weeks from last treatment to allow recovery from prior toxicity to a Grade 1 or less.
* The following exceptions are allowed: hormonal therapy - 1 week wash-out; radiation therapy - 3 week wash-out; weekly chemotherapy - 3 week wash-out
* Patients coming off experimental therapy with biological agents with long half lives (e.g., antibodies) not expected to cause myelotoxicity should be off treatment for at least 4 weeks.
* Negative serum pregnancy test within 14 days prior to the study entry and be practicing an effective form of contraception if hysterectomy and/or oophorectomy was not part of the prior treatment

Exclusion Criteria:

* Prior therapy with pegylated liposomal doxorubicin or doxorubicin.
* Prior therapy with BIBF 1120.
* Prior anti-angiogenic therapy with tyrosine kinase inhibitors (e.g. sorafenib, sunitinib, others). Note: Prior therapy with bevacizumab is allowed, provided that at least 3 months have elapsed since the last dose of bevacizumab.
* Grade 2 or greater neuropathy, at time of registration.
* Active cancer within the last 5 years, with the exception of superficial skin cancer (basal cell or squamous cell skin carcinoma), carcinoma in situ of the cervix, Stage I endometrial cancer with less than 50% invasion of the myometrium, or other adequately treated Stage I or II cancer in complete remission.
* Presence of active infection requiring antibiotic treatment, at time of registration.
* Presence of uncontrolled serious medical condition or psychiatric illness as determined by the treating physician, at time of registration.
* Known history of immune deficiency and be receiving combination anti-retroviral therapy
* Known or clinically manifest brain metastases, as progressive neurologic dysfunction may develop, that would confound the evaluation of neurologic and other adverse events.
* Presence of gastrointestinal disorders or abnormalities that would influence the absorption of the study drug.
* Presence of uncontrolled hypertension, arrhythmia, congestive heart failure or angina, at time of registration. Patients who have had a myocardial infarction or cardiac surgery should be at least 6 months from the event and free of active symptoms.
* Serious illness or concomitant non-oncological disease such as neurologic, psychiatric, infection disease or laboratory abnormality that may increase the risk associated with study participation or study drug administration.
* Major injuries within the past 4 weeks prior to start of study treatment with incomplete wound healing and/or planned surgery during the on-treatment study period.
* History of clinically significant hemorrhagic or thromboembolic event in the past 6 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2011-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Phase I: Safety and Toxicity of Treatment Regimen | 3 months
  To find the maximum tolerated dose (MTD) to be used during the Phase II trial and evaluate the safety and toxicity of the combination BIBF 1120 plus PLD in patients with recurrent or resistant epithelial ovarian or endometrial cancer.
Phase II: Objective Response Rate | 12 months
  To assess response rate (objective response) in patients with recurrent or resistant epithelial ovarian cancer treated with BIBF 1120 plus PLD.

SECONDARY OUTCOMES:
Phase I and II: Progression-Free Survival | 12 months
  To determine the progression-free survival of Phase I and II patients with recurrent or resistant epithelial ovarian cancer treated with BIBF 1120 plus PLD.
Phase I and II: Clinical Benefit | 12 months
  To determine the rate of clinical benefit for Phase I and II defined as:
  * the number of patients experiencing an objective response or
  * a CA125 response, in the absence of disease progression by clinical or radiographic criteria
  * sustained stable disease ≥ 3 months by clinical and radiographic criteria

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Matei, M.D., Principal Investigator — Hoosier Cancer Research Network
Locations (2):
- United States (2):
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - University of Wisconsin, Madison, Wisconsin

REFERENCES:
- [Background] Maria Creselda deLeon, Alesha Arnold, Emma Caroline Rossi, Jamie Case, Cynthia Johnson, Yan Zeng, Daniela Matei. Phase I trial of pegylated liposomal doxorubicin in combination with BIBF 1120 (nintedanib) in platinum-resistant ovarian cancer: Hoosier Oncology Group GYN10-149. J Clin Oncol 32:5s, 2014 (suppl; abstr 5541^)
- See also: Hoosier Oncology Group Homepage — http://www.hoosieroncologygroup.org